CLINICAL TRIAL: NCT03406741
Title: Neuropsychological Development and Functional Outcome Sin Children With Hirschsprung Disease at School Age - Hirschsprung
Brief Title: Neuropsychological Development and Functional Outcome Sin Children With Hirschsprung Disease at School Age
Acronym: Hirschsprung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-13; 2017-A01224-49 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hirschsprung's Disease (HD)
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child with Hirschsprung's disease (Experimental): Neuropsychological assessment at elementary school
  Interventions: Behavioral: psychometric evaluation; Behavioral: neuropsychological evaluation

INTERVENTIONS:
Behavioral: psychometric evaluation — Wechsler type composite scales (WISC)
Behavioral: neuropsychological evaluation — Evaluation of child behavior by the Goodman questionnaire: Strengths and Difficulties Questionnaire

SUMMARY:
Hirschsprung's disease (HD) is a rare congenital disease (1:5000) characterized by neonatal functional low bowel obstruction that is caused by aganglionosis of the distal bowel. HD treatment consists in surgery of colonic reduction in the early childhood, requiring afterward a long-term follow-up. In the long term complications (incontinence, constipation, enterocolitis, soiling)but also iterative anesthesia in childhood and repeated hospitalizations can have negative effects on child's development.

The main aim of the study is to estimate neuropsychological development at school age (6-10 years). Of children operated of HD Secondary aims are evaluation of the neuro-driving development and global health, comparison of quality of life levels to those of French population standards as well as to study the complex relations between on one hand the quality of life of these children and on the other hand the socio-demographic data, the initial clinical elements and the surgical coverage, as well as their health and current cognitive profile.

This multicenter study included pediatric surgery departments of Marseille. All children born between 1/1/2005 and 31/12/2010 and presenting HD represent the population. All the families will be contacted resting on the networks of set up follow-up. A written agreement will be collected with the parents. For all the participating children, a consultation will be organized: quality of life data (reported by children and by their parents in validated standardized questionnaires), clinical examination of the child, cognitive profile of the child. The duration of inclusion is scheduled for 12 months.

This is the first French study using auto-reported data on children's quality of life at school age affected by a HD. The results of this study will allow developing hypotheses on predictive risk factors for neuropsychological development disorders. Besides a better knowledge of the relation existing between these children quality of life and their functional results due to the disease could help clinicians in their medical reflections.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 8 to 13
* Child with Hirschsprung's disease (diagnosis confirmed by anatomopathological analysis),
* Child with no severe cerebral palsy
* Child with no developmental psychosis
* Child not showing amblyopia
* Child not deaf hearing
* Child able to answer a questionnaire in French language,
* a child whose parents or legal representatives have accepted the principle of participation in this study, and who have signed an informed consent,

Exclusion Criteria:

* Child deceased between birth and the date of assessment,
* Child with cerebral palsy
* Child whose parents or legal representatives refused to allow their child to participate in this study

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Evaluation of a sensory deficit | 12 months
  Administration d'un test psychometric de type Wechsler. The Wechsler Intelligence Scale for Children (WISC). The WISC-IV includes 15 subtests exploring four major components assessing the different intellectual skills essential to learning processes. The minimum score is 70, the normality between 90 ant 110, the maximum score is 130.

SECONDARY OUTCOMES:
Evaluation of child behavior by the Goodman questionnaire: Strengths and Difficulties Questionnaire (SDQ). | 12 months
  It includes 25 questions that are asked to parents. It is used within research, evaluating treatment outcome and as part of clinical assessment in order to examine a child's mental well-being. A total difficulties score is calculated using the SDQ, which ranges from 0-40. Each 1 point increase in the total difficulties score corresponds with an increase in the risk of developing a mental health disorder. Categories have been proposed by Youth in Mind authors in order to assess whether a child's score is close to average, slightly above average, high or very high.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No